CLINICAL TRIAL: NCT06305897
Title: Evaluation of the Tolerance (Main Objective) and Performance of Cyto-selective Difluoroethane-based Cryotherapy in the Treatment of Brown Spots (Solar and Senile Lentigines, Post-inflammatory Hyperpigmentation) on the Face
Acronym: CS5_10B
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cryonove Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CS5_10B
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Lentigo; Solar Lentigo; Post Inflammatory Hyperpigmentation
Keywords: cryotherapy; brown spots
MeSH Terms: conditions — Lentigo; Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Proof of concept study concerning 3 prototypes of cyto-selective cryotherapy devices corresponding to a modified CE marked medical device (ref: 822-v1).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Condition 1: (Experimental): Sequence of cryogenic gas (EC14_4osc)
  Interventions: Device: CRYONOVE (EC14_4osc)
- Condition 2: (Experimental): Sequence of cryogenic gas (EC+05_1osc)
  Interventions: Device: CRYONOVE (EC+05_1osc)
- Condition 3: (Experimental): Sequence of cryogenic gas (EC+05_2osc)
  Interventions: Device: CRYONOVE (EC+05_2osc)

INTERVENTIONS:
Device: CRYONOVE (EC14_4osc) — The prototype is a variant version from that of a CE marked MD already commercialized (Cryobeauty mains, Cryobeauty Pharma SAS, France) which produces a cryogenic spray sequence (EC14). The prototype is intended to treat pigmented spots of the face (PIH spots and senile and solar lentigos).
  Arms: Condition 1:
Device: CRYONOVE (EC+05_1osc) — The prototype is a variant version from that of a CE marked MD already commercialized (Cryobeauty mains, Cryobeauty Pharma SAS, France) which produces a cryogenic spray sequence (EC05_1osc). The prototype is intended to treat pigmented spots of the face (PIH spots and senile and solar lentigos).
  Arms: Condition 2:
Device: CRYONOVE (EC+05_2osc) — The prototype is a variant version from that of a CE marked MD already commercialized (Cryobeauty mains, Cryobeauty Pharma SAS, France) which produces a cryogenic spray sequence (EC05_2osc). The prototype is intended to treat pigmented spots of the face (PIH spots and senile and solar lentigos).
  Arms: Condition 3:

SUMMARY:
The goal of this clinical trial is to compare the 3 different prototype of cyto-selective cryotherapy devices (name of the devices : CRYONOVE) use in brown spots on the face of subject from different ethnicities. The main questions it aims to answer are:

* the tolerance of 3 prototypes of cyto-selective cryotherapy treatments
* the performance of 3 prototypes of cyto-selective cryotherapy treatments

Participants will be treated for each spots with a definied prototype during 6 treatment visits.

Researchers will compare the tolerance and performance of the 3 prototypes.

ELIGIBILITY:
Inclusion Criteria:

1. Subject having signed a written informed consent form (ICF) to participate in the investigation obtained according to ISO 14155:2020 - Good Clinical Practice (GCP);
2. Healthy male and female subjects, 18 to 75 years old (inclusive), and Fitzpatrick's skin type (II-VI) (1);
3. Subject of Caucasian and or melanin-rich ethnicity skins;
4. Subject presenting at least two brown spots on the face with ≥ 3 and ≤ 6 mm in diameter;
5. Female subject of non-childbearing potential, defined as woman without uterus and/or both ovaries, surgically sterile (at least 6 months prior to Screening visit) or post-menopausal (at least one year post cessation of menses);
6. Female subject of childbearing potential who has been, in the opinion of the Investigator, using an approved method of birth control for at least 1 month prior to Screening visit and agreeing to continue adequate contraception during the entire study period;

   Reliable methods of contraception are:
   * hormonal methods or intrauterine device in use since at least 1 month prior to Screening visit and during the investigation period;
   * bilateral tubal ligation since at least 3 months prior to Screening visit and during the investigation period;
   * barrier methods in use at least 14 days prior to Screening visit;
   * vasectomized partner;
   * sexual abstinence defined as refraining from heterosexual intercourse for at least 3 months prior to Screening visit and during the entire period of risk associated with the study products.
7. Subject who has not been exposed to UV within at least two months prior to the screening visit and agreeing to avoid exposure to UV radiation (tanning beds, phototherapy and sunlight) for the whole study duration;
8. Subject able to comprehend the full nature and the purpose of the investigation, including possible risks and side effects, and subjects able to cooperate with the Investigator and to comply with the requirements of the entire investigation (including ability to attend all the planned investigation visits according to the time limits), based on Investigator's judgement;
9. Subject affiliated to a health social security system (according to French Law).

Exclusion Criteria:

1. Female subject who is pregnant, parturient or breast feeding;
2. Female subject of childbearing potential having a positive urinary pregnancy test at Day 0;
3. Subject having performed cosmetic treatments (e.g., exfoliants, scrubs or selftanners, facial UV) in the month before the start of the study on the face (see restrictions paragraph);
4. Subject having performed cosmetic or aesthetic treatments by a dermatologist (e.g., laser, IPL, peeling, creams, cryotherapy) in the last 6 months on the face;
5. Subject receiving systemic or local treatment (e.g., dermocorticoids, corticosteroids, diuretics) likely to interfere with the evaluation of the parameter studied;
6. Subject affected by dermatosis, autoimmune disease, systemic, chronic or acute disease, or any other pathology that may interfere with treatment or influence the results of the study (e.g., people with diabetes or circulatory problems, allergic to cold, Raynaud's syndrome);
7. Subject with clinically significant skin condition on the tested area (e.g., active eczema, psoriasis, rosacea, scleroderma, acne, dermatitis) or presence on the tested area of skin lesions, scars, tattoos;
8. Concomitant participation in other clinical trials/investigations or participation in the evaluation of any IMD/IP during 2 months before this study;
9. Protected subject as defined in the Articles of the French Public Health Code: Article 1121-7: person deprived of liberty by a judicial or administrative decision, or subject to psychiatric care or person admitted to a health or social institution for purposes other than the research. Article 1121-8: adult person subject to a legal protection measure or unable to express his/her consent;
10. Subject unable to communicate or cooperate with the Investigator due to poor mental development, language problems or impaired cerebral function;
11. Subject currently participating in another clinical study or being in an exclusion period of another clinical study;
12. Subject having received 6000 euros indemnities for participation in clinical trials/investigations in the 12 previous months, including participation in the present study (according to French Law).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Tolerance | Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70, Day 84
  The primary objective of this clinical investigation is to evaluate the tolerance (IGA scale) of 3 prototypes of cyto-selective cryotherapy treatments applied on the brown spots on the face of subject from different ethnicities (Caucasian and melanin-rich skins). A brown spot is defined as solar or senile lentigo (SSL) and post-inflammatory hyperpigmentation (PIH).
  -> IGA Scale : Investigator's Global Assessment - 6 points - Scale in 6 points (0 to 5) 0 = clear of hyperpigmentation
  1. = almost clear of hyperpigmentation
  2. = mild, but noticeable hyperpigmentation
  3. = moderate hyperpigmentation (medium brown in quality)
  4. = severe hyperpigmentation (dark brown in quality)
  5. = very severe hyperpigmentation (very dark brown, almost black in quality)

SECONDARY OUTCOMES:
Performance | Day 7, Day 14, Day 21, Day 28, Day 35, Day 42, Day 56, Day 70, Day 84
  The secondary objective of this clinical investigation is to evaluate the performance of 3 prototypes of cyto-selective cryotherapy treatments applied on the brown spots on the face of subject from different ethnicities (Caucasian and melanin-rich skins).
  * Standardized photographs will be taken before the treatment at each visit (C-cube).
  * Color Chart (color and lightness) only for Caucasian skins.

IPD SHARING:
Plan to Share IPD: No